CLINICAL TRIAL: NCT06438419
Title: Parkinsonism-Related Oscillations in the Cortico-Basal Ganglia-Thalamic Network During Movement: Beyond the Frequency Range
Acronym: MOVOSCILLCBGT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Université de Bordeaux, IMN, UMR CNRS 5293 (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CHUBX 2023/63
Record Dates: First submitted 2024-05-27; First posted 2024-05-31 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Parkinson Disease; Hyperkinesis; Hypokinesia
Keywords: Parkinson disease; hypokinetic disorders; dyskinesia; networks; basal ganglia
MeSH Terms: conditions — Parkinson Disease; Hyperkinesis; Hypokinesia; Dyskinesias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Recruited patient (Experimental): Patient with idiopathic Parkinson's disease and having a STN DBS with a PERCEPT™ for less than a year or being candidate for subthalamic nucleus deep brain stimulation with the PERCEPT™ device (first-implantation)
  Interventions: Other: Electrophysiological recordings

INTERVENTIONS:
Other: Electrophysiological recordings — Electrophysiological recordings will be made during a motor task in four different conditions:
  1. without pharmacological treatment and without stimulation (Off condition),
  2. without pharmacological treatment and during stimulation (DBS condition),
  3. during pharmacological treatment and without stimulation (DOPA condition),
  4. during pharmacological treatment and stimulation (DOPA+DBS condition).

SUMMARY:
Expression of hypokinetic and hyperkinetic motor symptoms in Parkinson's disease (PD) is associated with pathological synchronous oscillations of neuronal activity (local field potential/LFP) in the cortico-subcortical network with a wide frequency range. In the present project, we propose to study cortico-subcortical oscillations and their synchronization in patients operated for PD (subthalamic deep brain stimulation (STN-DBS)) during distinct pharmacological and stimulation conditions (hypokinetic and hyperkinetic), using a simple motor task.

DETAILED DESCRIPTION:
To define the link between the characteristics of neuronal oscillations (frequency, amplitude, phase relationship) within the cortico-subcortical network and the movement, we designed a simple motor task of gripping/pulling a lever. The LFPs will be collected at the cortical and subcortical levels (STN) during the motor task using a high-resolution EEG (HR-EEG) and the Percept™ system (Medtronic). Recordings will be realized in four conditions: without pharmacological treatment and without stimulation (Off condition), without pharmacological treatment and during stimulation (DBS condition), during pharmacological treatment and without stimulation (DOPA condition) and during pharmacological treatment and stimulation (DOPA+DBS condition).

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* 18 to 75 years-old
* With idiopathic Parkinson's disease
* Having a STN-DBS with a PERCEPT™ for less than a year or being candidate for STN-DBS with the PERCEPT™ device (first-implantation)
* Able to perform the simple motor task
* Patients covered by a health insurance scheme
* Giving free, informed, written consent signed by the participant and the investigator.

Exclusion Criteria:

* Be incapable of giving consent personally.
* Be subject to a legal protection measure (curatorship, guardianship) or be placed under judicial protection.
* Being pregnant or breastfeeding
* Present a serious and/or decompensated somatic or psychiatric illness.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-16 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Cortico-subcortical electrophysiological coherence | At inclusion (Day 0)
  Statistically significant difference in the cortico-subcortical electrophysiological coherence value between a movement performed in hypokinetic condition and a movement performed in hyperkinetic condition

SECONDARY OUTCOMES:
Spectral signal power | At inclusion (Day 0)
  Demonstration of a significant difference in spectral signal power between movement in hypokinetic and hyperkinetic conditions.
Effect of STN-DBS on spectral signal power | At inclusion (Day 0)
  Demonstration of a significant effect of STN-DBS on spectral signal power and cortico-subcortical synchronization during movement in hypokinetic or hyperkinetic conditions
Correlation between semiological characteristics | At inclusion (Day 0)
  Demonstration of a statistical correlation between semiological characteristics (hypo- and hyperkinesia, movement parameters (reaction time and movement time)) and electrophysiological characteristics.

CONTACTS AND LOCATIONS:
Locations (1):
- Bordeaux University Hospital, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No